CLINICAL TRIAL: NCT02501174
Title: Study of Elderly Patients With Cancer and Seen in Consultation of Geriatric Oncology in the Nord Pas-de-Calais (CONSOG).
Status: Completed | Type: Observational
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Other Study IDs: CONSOG-1401
Record Dates: First submitted 2015-07-02; First posted 2015-07-17 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Cancer
Keywords: Geriatric oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to establish a common geriatric oncology medical database. The patients concerned are the patients having benefited from a geriatric oncology consultation in one of the participating centres. This database is designed with a view on the one hand to better describe to better understand this population and on the other hand to facilitate the conduct of future retrospective or prospective studies on this population. The constitution of this observatory of patients seen in consultation should facilitate the development of studies from the analysis of data collected, and occasional surveys by the rapid identification of cases. Data from this database could provide clinicians with valuable informative elements of descriptive epidemiology and concerning the organization of care in the geriatric oncology field.

DETAILED DESCRIPTION:
The study is presented during the first consultation of oncogeriatric care or after this consultation (for patients having benefited from the consultation between January 2014 and October 2014) : the patient is informed with an information note and is told that he can express its opposition to the use of its clinical data. In case of no opposition from the patient, the referent geriatrician will complete the patient form with the requested data and will forward it for computerized processing.

ELIGIBILITY:
Inclusion Criteria:

* Patient seen in consultation of geriatric oncology in one of the participating centres in Nord Pas-de-Calais.
* Age ≥ 65 years
* Patient having been informed and not opposing the computerized processing of its data.

Exclusion Criteria:

* Patient having opposed the use of its medical data.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients included are patients followed in one of the participating centres and not opposing the use of their medical data.
Sampling Method: Non-Probability Sample
Enrollment: 2914 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Measurement of the prevalence of different clinical criteria of interest : demographic characteristics, disease state, patient status according to the geriatric criteria (Comprehensive Geriatric Assessment (CGA)). | Up to 5 years

SECONDARY OUTCOMES:
Measurement of the prevalence of different medical and social criteria of interest. | Up to 5 years
  Patient's life characteristics (place of living, isolation) and the helps set up (presence of a natural caregiver, sources of professional help).
Measurement of the association between one or more factors of interest (clinical, biological and medical and social) related to a proposal to amend or not the initially proposed therapeutic strategy. | Up to 5 years
Percentage of patients included in trials. | Up to 5 years
Temporal evolutions of clinical, medical and social characteristics. | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Cédric GAXATTE, MD, Principal Investigator — CHRU de Lille
Locations (15):
- France (15):
  - Centre Hospitalier d'Arras, Arras
  - Centre Hospitalier, Béthune
  - Centre Hospitalier, Boulogne-sur-Mer
  - Centre Hospitalier, Douai, Douai
  - Centre Hospitalier, Dunkirk
  - Hospitalier Le Cateau-Cambresis, Le Cateau-Cambrésis
  - Polyclinique de Riaumont, Liévin
  - CHRU de Lille, Lille
  - Hôpital Saint Vincent de Paul, Lille
  - Centre Oscar Lambret, Lille
  - Hôpital Saint-Philibert, Lomme
  - Clinique Saint Jean, Roubaix, Roubaix
  - Centre Hospitalier, Tourcoing
  - Centre de cancérologie Les Dentellières, Valenciennes
  - Centre Hospitalier, Valenciennes

IPD SHARING:
Plan to Share IPD: No